CLINICAL TRIAL: NCT03305367
Title: Dose-response Effect of Pine Nut Oil as a Dual FFA1 and FFA4 Agonist on Glucose Tolerance, Incretins, Appetite and Tolerability in Healthy Humans.
Brief Title: Dose-response Effect of Pine Nut Oil as a Dual FFA1 and FFA4 Agonist on Glucose Tolerance in Healthy Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Karina Vejrum Sørensen, MSc, PhD-student, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PINO3
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Subjects complete three oral glucose tolerance tests (OGTT) on different days, with a minimum of one week in between. First visit is a combined screening and baseline OGTT, with no supplementation. At the second and third visit subjects are randomly assigned to either 3 g of hydrolyzed pine nut oil or 6 g of hydrolyzed pine nut oil.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Screening/Baseline (No Intervention): A standard OGTT with no supplementation/intervention
- Hydrolyzed pine nut oil low dose (Experimental): Standard OGTT supplemented with 3 g of hydrolyzed pine nut oil
  Interventions: Dietary Supplement: Hydrolyzed pine nut oil
- Hydrolyzed pine nut oil high dose (Experimental): Standard OGTT supplemented with 6 g of hydrolyzed pine nut oil
  Interventions: Dietary Supplement: Hydrolyzed pine nut oil

INTERVENTIONS:
Dietary Supplement: Hydrolyzed pine nut oil — Randomized cros-over intervention of 3 OGTT with no oil, low dose or high dose.
  Arms: Hydrolyzed pine nut oil high dose; Hydrolyzed pine nut oil low dose

SUMMARY:
Several free fatty acids receptors (FFARs) have been discovered. These have been implicated in metabolic processes and inflammation. Consequently, these receptors have attracted interest as targets for the treatment of metabolic and inflammatory diseases, including obesity and type 2 diabetes. Two of these FFARs (FFA1, FFA4), which is activated by specific free fatty acids (FFAs), is expressed on enteroendocrine cells, pancreatic beta-cells and adipocytes. They have been linked to 1) increased glucagon-like peptide-1 (GLP-1) secretion and hence the incretin-mediated increase in glucose-stimulated insulin secretion (GSIS) and suppression of glucagon secretion, 2) a direct positive effect on GSIS, 3) reduced inflammation and 4) improved insulin sensitivity. These functions and the abundance of fatty acids in food suggest that FFARs can be considered as nutrient sensing regulators of metabolism. Roux-en-Y gastric bypass (RYGB), frequently results in immediate beneficial effects on glucose metabolism and often complete remission of type 2 diabetes. This may in part be explained by increased GLP-1 levels after surgery. It appears that the effect depends on nutrient delivery directly to the lower parts of the small intestine. It is possible that the RYGB effects are partly due to enteroendocrine stimulation of FFA1 and perhaps FFA4 by direct nutrient delivery, i.e. FFA release in the lower intestines. Pinolenic acid from pine nuts has been shown to be a potent dual FFA1/FFA4 agonist.

Based on these findings the investigators have planned a number of human intervention studies in order to investigate 1) the optimal oral formulation of pine nut oil 2) whether it is possible to mimic the beneficial effects observed after RYGB, 2) if it is possible to increase GLP-1 secretion by stimulating FFA1/FFA4 on enteroendocrine cells causing improved GSIS and increased satiety and 3) enhancement of GSIS by directly stimulating FFA1 on beta-cells.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is one of the greatest health challenges worldwide. The disease is strongly associated with obesity, and develops via pre-diabetic conditions, where insulin resistance and low-grade inflammation play an important role, to T2D, where failure of the pancreatic beta-cell to compensate for insulin resistance causes hyperglycemia. According to recent estimates, 350 million people worldwide suffer from diabetes. The disease typically leads to many years of reduced quality of life due to complications such as cardiovascular disease (CVD), blindness, kidney failure and amputations. T2D is estimated to be the 4th leading cause of death in the Western world with 5-10 years reduced life expectancy. It is generally agreed that a healthy diet and increased physical activity are effective in preventing T2D, and also may help to achieve a better control of T2D and reduce the risk of CVD. There is, however, not a general agreement as to what a healthy diet constitutes.

During the last decade, several cell surface receptors that respond to free fatty acids (FFAs) have been discovered. These free fatty acid receptors (FFARs) belong to the superfamily of G protein-coupled 7-transmembrane receptors (GPRs), and have all been implicated in metabolic processes, energy expenditure and inflammation. Consequently, several of the receptors have attracted interest as potential targets for the treatment of metabolic and inflammatory diseases, including obesity and T2D.

FFA1 (GPR40), which is activated by long-chain FFAs, is highly expressed in pancreatic β-cells and increases glucose-stimulated insulin secretion (GSIS) [4]. There is evidence that FFA1 is also expressed in intestinal enteroendocrine cells, where it promotes secretion of incretin hormones such as GLP-1 and glucose-dependent insulinotropic peptide (GIP). GLP-1 is highly interesting for treatment of obesity and T2D because of its ability to increase GSIS, enhance β-cell growth, increase insulin sensitivity, reduce gastric motility, increase satiety and cause a loss of weight. The published phase II clinical trial with the selective FFA1 agonist TAK-875 demonstrated high efficacy in reducing plasma glucose without increased incidence of hypoglycemia, and has caused considerable interest in the receptor as a new target for treatment of T2D.

FFA4 (GPR120), which is activated by unsaturated long-chain FFA, is expressed in the gastrointestinal system, adipose tissue, and β-cells, and is reported to promote GLP-1 secretion from intestinal cells, to counteract inflammation and to increase insulin sensitivity in adipose tissue. Notably, dysfunctional FFA4 was recently connected to the development of obesity in both mice and humans. This has considerably increased the interest on the receptor as a target for obesity and metabolic diseases. This is supported by indications that unsaturated FFAs revert diet-induced hypothalamic inflammation through FFA4, and thereby reduce body weight in diet-induced obese mice. These FFARs are thus expressed in different tissues in the body where they potentially can affect metabolic and inflammatory conditions such as T2D and obesity.

These functions combined and the abundance of fatty acids in food suggests that FFARs can be considered as nutrient sensing regulators of metabolism.

Roux-en-Y gastric bypass (RYGB) surgery, often used to treat severe obesity, frequently results in immediate beneficial effects on glucose metabolism in T2D, often with complete remission. These effects are in part independent of weight loss, but may be explained by a significant increase in GLP-1 levels immediately after surgery. Thus, it appears that the effect depends on delivery of nutrients and pancreatic juices directly to the lower parts of the ileum. Normally, FFAs are rapidly absorbed in the upper parts of the gastrointestinal tract. It is therefore possible that the RYGB effects are partly due to enteroendocrine stimulation of FFA1 and perhaps FFA4 by direct nutrient delivery that is FFA release in the lower intestines. A hypothesis to be investigated in this PhD project is that delivery of a specific naturally occurring polyunsaturated FFA with proven high efficacy on both FFA1 and FFA4 directly to the lower intestines can mimic the beneficial effects observed after RYGB with less expense and fewer adverse effects.

Delivery of a higher load of unabsorbed FFA to the distal small intestine can be achieved by taking advantage of enteric coating that dissolves at pH >6.0, which is observed in the lumen of the distal jejunum, ileum and colon, and is independent of the colonic flora. This enteric coating technology is well established for delivering drugs to the ileum and colon. The potential positive effect of this principle was recently reported in a small cohort of patients with T2D. Thus, delivery of small amounts of lauric acid (a C12 fatty acid) to the distal gut using enteric-coated pellets stimulated GLP-1 secretion and lowered postprandial glucose levels in response to meals. No chronic effects where tested in this study. Although not suggested by the authors, the increased release of GLP-1 could involve direct stimulation of FFAR1 and/or FFAR4 by lauric acid in the distal gut.

As a part of the FFARMED project supported by the Danish Council for Strategic Research, a screening of 36 relevant FFAs and their ability to act as FFA1 and FFA4 agonists in vitro have been carried out to identify the most potent naturally occurring dual FFA1/FFA4 agonist for clinical studies. Of these, the polyunsaturated fatty acid (PUFA), pinolenic acid showed a significantly higher efficacy than the others, and was therefore selected for further studies. To further support this choice, the effect of pinolenic acid has been tested using a small dose (100 mg/kg) given 30 min prior to an oral glucose tolerance test in mice. Convincingly, purified pinolenic acid significantly improved glucose tolerance by reducing glucose levels when compared to control (corn oil). The efficacy was similar to that obtained with a pharmaceutical selective FFA1 agonist (TUG-905). Pinolenic acid is a fatty acid contained in Siberian Pine nuts, Korean Pine nuts and the seeds of other pines. The highest percentage of pinolenic acid (~20%) is found in Siberian Pine nuts and the oil produced from them. Korean Pine nut oil given as hydrolyzed FFAs, but not as triglycerides has been reported to increase secretion of GLP-1 and decrease appetite in overweight females. This is in coherence with previous results in mice, and indicates that purified pinolenic acid may be superior in improving glucose metabolism.

Hypotheses: As described, the expression of FFA1 and FFA4 on intestinal enteroendocrine cells, pancreatic beta-cells and adipose tissue has been linked to 1) increased secretion of GLP-1 and hence the incretin-mediated increase in GSIS and suppression of glucagon secretion, 2) a direct positive effect on GSIS, 3) reduced inflammation and 4) improved insulin sensitivity. Based on the above findings, the investigators are performing a number of clinical trials using pinolenic acid derived from Siberian pine nuts as a naturally occurring dual FFA1/FFA4 agonist. The investigators hypothesize that ingestion of a small amount of pinolenic acid given as enteric-coated pellets dissolved in the lower intestines will 1) increase GLP-1 secretion by stimulating FFA1/FFA4 on enteroendocrine cells causing improved GSIS and increased satiety, 2) enhance GSIS by directly stimulating FFA1 on beta-cells, and 3) attenuate the low-grade inflammation seen in insulin resistant conditions such as obesity and T2D by stimulating FFA4 on adipocytes.

The aim of this study is to investigate: The dose-response effect of delayed release pinolenic acid (hydrolyzed pine nut oil) on glucose tolerance, insulin and incretin secretion, appetite and tolerability in healthy humans.

This registration covers the third off five planned pilot studies investigating the effect of hydrolyzed pine nut oil on glucose metabolism during an oral glucose tolerance test.

ELIGIBILITY:
Inclusion criteria: body mass index of 27.5-40 kg/m2 and age between 40-70 years. Healthy subjects, non-smoking, without a close relative history of diabetes, no usage of prescription drugs or dietary supplements within the past month (birth control allowed). Subjects should be able to give informed consent and have no trouble swallowing capsules.

Exclusion criteria: impaired glucose tolerance measured as two hours OGTT glucose concentration above 7.7 mmol/l, abnormal screening blood samples, food allergies, more than 3kg weight change or restrictive dieting two months prior, severe hypertension or history of gastrointestinal disease or surgery.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 4 hours OGTT
  Area under the curve of blood glucose
Insulin and C-peptide | 4 hours OGTT
  Area under the curve of Insulin and C-peptide
Incretins | 4 hours OGTT
  Area under the curve of incretins
ghrelin | 4 hours OGTT
  Area under the curve of ghrelin
appetite | 4 hours OGTT
  Visual analog scale - area under the curve
Gastrointestinal tolerability | 4 hours OGTT
  Visual analog scale -mm

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Højlund, MD, Principal Investigator — Department of Endocrinology
Locations (1):
- Department of Endocrinology, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
Not intended at the moment

REFERENCES:
- [Derived] Sorensen KV, Korfitzen SS, Kaspersen MH, Ulven ER, Ekberg JH, Bauer-Brandl A, Ulven T, Hojlund K. Acute effects of delayed-release hydrolyzed pine nut oil on glucose tolerance, incretins, ghrelin and appetite in healthy humans. Clin Nutr. 2021 Apr;40(4):2169-2179. doi: 10.1016/j.clnu.2020.09.043. Epub 2020 Oct 2. PMID 33059911